CLINICAL TRIAL: NCT03891433
Title: Piperacillin/Tazobactam Versus Carbapenems in Non-bacteremic Urinary Tract Infections Due to Extended-spectrum Β-lactamase (ESBL)-producing Escherichia Coli or Klebsiella Pneumoniae - (CAPITIS Study)
Brief Title: Piperacillin/Tazobactam Versus Carbapenems in Non-bacteremic UTI Due to -ESBL-producing Enterobacteriaceae
Acronym: CAPITIS
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Low admission of patients with the condition to the hospital because it is a reference center for care of the SARS-CoV-2 pandemic
Sponsor: Universidad del Norte (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUN-INF-CAPITIS-2018-1
Record Dates: First submitted 2019-03-11; First posted 2019-03-27 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Urinary Tract Infections; Enterobacteriaceae Infections; Infection Due to ESBL Bacteria; Carbapenem; Escherichia Coli Infection; Klebsiella Pneumoniae Infection; Clinical Trial; Drug Resistance, Bacterial
Keywords: adult; Equivalence Trial; Randomized Controlled Trial; Comparative Study; Anti-Bacterial Agents/therapeutic use*; Meropenem; Ertapenem; Piperacillin, Tazobactam Drug Combination; Escherichia coli Infections/drug therapy; Klebsiella Infections/drug therapy
MeSH Terms: conditions — Urinary Tract Infections; Enterobacteriaceae Infections; Escherichia coli Infections | interventions — Meropenem; Ertapenem; Piperacillin; Tazobactam; Solutions; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An investigator of the research project conducted daily monitoring of the patient and will not be involved in clinical decisions. The statistical analyzes performed finally be blind to the treatment received by the patients (carbapenems vs piperacillin/tazobactam).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbapenems group (Active Comparator): Meropenem (1g intravenously every 8 hours or adjusted to renal function) or Ertapenem (1g intravenously every 24 hours or adjusted to renal function) by 10 days.
  Interventions: Drug: Meropenem; Drug: Ertapenem 1000 MG
- Piperacillin/tazobactam. (Active Comparator): Piperacillin / Tazobactam (4.5gr intravenously every 6 hours or adjusted to renal function) by 10 days.
  Interventions: Drug: Piperacillin, Tazobactam 4-0.5G Solution for Injection

INTERVENTIONS:
Drug: Meropenem — Carbapenems group intervention.
  Arms: Carbapenems group
Drug: Ertapenem 1000 MG — Carbapenems group intervention.
  Arms: Carbapenems group
Drug: Piperacillin, Tazobactam 4-0.5G Solution for Injection — Piperacillin/Tazobactam group intervention.
  Arms: Piperacillin/tazobactam.

SUMMARY:
This study evaluates the efficacy in achieving clinical cure in non-bacteremic urinary tract infections (UTI) caused by Escherichia coli or Klebsiella pneumoniae producers of extended-spectrum β-lactamases (ESBL) in adult patients. Half of participants will receive Piperacillin/Tazobactam as treatment, while the other half will receive Carbapenems.

The investigators will verify that Piperacillin/Tazobactam is not inferior in achieving clinical cure, and that is not associated with a higher risk of adverse events in the directed treatment of non-bacteremic UTI compared to Carbapenems.

The researchers hope to improve the use of antibiotics in the non-bacteremic UTI, reducing the "collateral damage" related to a deterioration in the prognosis of patients and the generation of resistant germs caused by the use of broad-spectrum antibiotics as carbapenems.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is a common cause of hospitalization worldwide, the prevalence throughout the life of UTI has been reported in about 50,000 cases per 100,000 women and 13,000 per 100,000 men in the United States. Hospitalization for community-acquired UTI is about 33%. Furthermore, the UTI related to bladder catheterization during hospitalization is the most common type of infection acquired, representing 40% of all nosocomial infections. UTI hospitalization is associated with a high cost to the healthcare system.

The diagnosis of UTI is based on demonstrating the presence of bacteria urine in patients with suggestive clinical manifestations and verifying the host's inflammatory response to infection. The most common etiological agents include Escherichia coli, Klebsiella spp, and Proteus spp, with different prevalence and antibiotic susceptibility profiles among different populations.

Currently the appropriate treatment of UTI is a growing concern in the medical community because Gram-negative, specifically Enterobacteriaceae, bacteria have acquired genes encoding antibiotic resistance mechanisms. The β-lactamase spread spectrum (ESBL) are documented with increasing frequency among microorganisms causing UTI. Current treatment options for ESBL bacteria include nitrofurantoin, fosfomycin, piperacillin-tazobactam, carbapenems, and aminoglycosides.

Carbapenems and piperacillin-tazobactam are antibiotics used in medical practice for many years, both therapies are licensed for the treatment of non-bacteremic UTI; however, so far there is not enough evidence to discriminate the best choice for the treatment of non-bacteremic UTI (although carbapenems are considered drugs of choice for infections caused by these microorganisms), but carbapenems use has been associated with an increased risk of "collateral damage" related to the generation of resistant germs.

The investigators will compare between piperacillin/tazobactam and carbapenems the effectiveness in achieving clinical cure for non-bacteremic UTI caused by ESBL microorganisms. Researchers principal hypothesis is that Piperacillin/tazobactam is not inferior to carbapenems in achieving clinical cure in the targeted treatment of UTI caused by non-bacteremic due to E. coli or K. pneumoniae ESBL in adults requiring hospitalization. Researchers will verify too if Piperacillin/Tazobactam is not associated with increased risk of adverse events during the targeted treatment of non-bacteremic ITU caused by E. coli or K. pneumoniae ESBL in adults requiring hospital admission, compared with Carbapenems therapy.

To perform the protocol researchers follows the recommendations for the design of trials investigating treatment options for resistant bacteria multidrug (Uncomplicated Urinary Tract Infections: Developing Drugs for Treatment) of the United States Agency for Food and Drug Administration (FDA).

Participants will be included in the study with informed consent. The study variables will be obtained by patient interview and review of medical history. Variables will be recorded in a computerized database developed specifically for this study, with exclusive access for the researchers.

The estimated project duration is 2 years expected to begin in april of 2019.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with hospital admission for non-bacteremic UTI caused by E. coli or K. pneumoniae ESBL susceptible to piperacillin/tazobactam and carbapenems.
* Presence of any risk factor associated with UTI due to ESBL germs: older age 64 years, diabetes mellitus, bladder catheter, previous antibiotics in the last 6 months, hospitalization in the last 6 months, urological surgery in the last 30 days, infections recurrent urinary.
* Diagnosis of UTI confirmed by: 1) fever, 2) urine culture> 100000 CFU with isolation E. coli or K. pneumoniae ESBL susceptible to piperacillin / tazobactam and carbapenems, and 3) lumbar and / or abdominal pain with or without low urinary symptoms (dysuria, tenesmus, urgency), and 4) no other cause that explains the patient's symptoms
* Signed informed consent.
* Negative pregnancy test in fertile women.

Exclusion Criteria:

* Non-acceptance of participation in the study.
* Pregnancy.
* Hypersensitivity and/or previous intolerance to penicillins, piperacillin/tazobactam or carbapenems.
* Bacteremia, hematogenous infection or other concomitant infection.
* Immunosuppression.
* In case of obstructive uropathy, lack of early surgical resolution.
* Evidence of acute or chronic prostatitis.
* Renal abscess
* Polycystic disease in the kidneys.
* Palliative care or life expectancy <90 days.
* Heart failure (NYHA) functional class III or IV.
* Liver cirrhosis.
* Renal insufficiency in dialysis treatment.
* Empirical active treatment against bacteria isolated by urine cultures other than E. coli or K. pneumoniae BLEE.
* Participation in another clinical trial for infections.
* Hypersensitivity to amide-type local anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Clinical cure. | At 5-7 day after the end of treatment (cure test), or for early response after 5 days from the start of treatment.
  Complete resolution of non-bacteremic urinary tract infection signs or symptoms (dysuria, urinary frequency, urinary urgency, suprapubic pain or temperature greater than 38 degrees Celsius) present at trial entry (and no new signs or symptoms) until the duration of investigational antibacterial drug therapy.
  Investigators will compare the rate of clinical cure between the two treatment lines.

SECONDARY OUTCOMES:
Microbiologic cure. | At the 5-7 day after the end of treatment (cure test).
  Clinical cure (primary outcome) and demonstration that the bacterial pathogen found at trial entry is reduced to fewer than 100.000 CFU/mL on control urine culture.
  Investigators will compare the rate of microbiologic cure between the two treatment lines.
Mortality in patient follow-up. | Until day 30 after the first day of administration of the study drugs.
  All-cause Mortality Rate in the CAPITIS Study Population (Piperacillin/Tazobactam Versus Carbapenems in Non-bacteremic Urinary Tract Infections Due to Extended-spectrum β-lactamase (ESBL)-Producing Escherichia Coli or Klebsiella Pneumoniae.
Length of hospital stay in patient follow-up. | Until day 30 after the first day of administration of the study drugs.
  Time since the assignment of the randomization until the patient leaves the hospital.
Relapse. | Daily until day 30 after the first day of administration of the study drugs.
  Proportion of Subjects in the CAPITIS Study Population with a Relapse (All Indications).
  Development of non-bacteremic urinary tract infection signs or symptoms (dysuria, urinary frequency, urinary urgency, suprapubic pain or temperature greater than 38 degrees Celsius) in patients with previous clinical and microbiological cure, plus positive urine culture with the same microorganism isolated in initial culture.
  Investigators will compare the risk of relapse with each regimen.
Reinfection. | Daily until day 30 after the first day of administration of the study drugs.
  Proportion of Subjects in the CAPITIS Study Population With a Reinfection (All Indications).
  Development of non-bacteremic urinary tract infection signs or symptoms (dysuria, urinary frequency, urinary urgency, suprapubic pain or temperature greater than 38 degrees Celsius) in patients with previous clinical and microbiological cure, plus positive urine culture with different strains isolated in initial culture.
  Investigators will compare the risk of reinfection with each regimen.
Resistant clinical isolates in patient follow-up. | Daily until day 30 after the first day of administration of the study drugs.
  Proportion of Subjects in the CAPITIS Study Population With Resistant clinical isolates.
  Appearance of clinical isolates of Escherichia coli or Klebsiella pneumoniae resistant piperacillin/tazobactam or carbapenems demonstrated in urine cultures will be evaluated.
Adverse events in patient follow-up. | Daily until day 30 after the first day of administration of the study drugs.
  Proportion of Subjects in the CAPITIS Study Population With Adverse events (All Indications).
  Any related adverse event occurring from the signing the informed consent form to end of follow.
  Investigators have created a data collection notebook, a daily follow-up will be made in the participants and adverse events in patient will be recorded.
ICU admission in patient follow-up. | Daily until day 30 after the first day of administration of the study drugs.
  Proportion of Subjects in the CAPITIS Study Population With ICU admission (All Indications).
  Any admission to intensive care unit occurs from signing the informed consent form to end of patient follow.
  Investigators have created a data collection notebook, a daily follow-up will be made in the participants and all admission in ICU will be recorded.
Clinical or microbiological failure of antibiotic therapy in patient follow-up. | Daily until day 30 after the first day of administration of the study drugs.
  Proportion of Subjects in the CAPITIS Study Population With Clinical or microbiological failure of antibiotic therapy (All Indications).
  Failure to achieve clinical or microbiologic cure until day 30, or die at any time since signing the informed consent form to end of follow-up.
  Authors defined the clinical therapeutic failure as the persistence of at least one urinary symptom in the patient at the time of follow-up despite antibiotic therapy. Microbiological failure has been defined as the persistence of bacteria isolation major to 10.000 UFC/ml in second urine culture carried out in the study participant despite antibiotic therapy.
  Investigators have created a questionnaire which will be checked daily with a urinary symptoms list. All findings will be recorded in a data collection notebook.

CONTACTS AND LOCATIONS:
Overall Officials: Diego F Viasus Perez, MD. PhD., Principal Investigator — Universidad del Norte´s Hospital-Infectious Diseases.; Andres F Estupinan Bohorquez, MD, Principal Investigator — Universidad del Norte
Locations (1):
- Universidad del Norte´s Hospital, Soledad, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Hwang K. Semiquinone of D-amino acid oxidase. Med J Osaka Univ. 1967 Dec;18(3):175-84. No abstract available. PMID 4386243
- [Background] Pitout JD, Laupland KB. Extended-spectrum beta-lactamase-producing Enterobacteriaceae: an emerging public-health concern. Lancet Infect Dis. 2008 Mar;8(3):159-66. doi: 10.1016/S1473-3099(08)70041-0. PMID 18291338
- [Background] Paterson DL, Bonomo RA. Extended-spectrum beta-lactamases: a clinical update. Clin Microbiol Rev. 2005 Oct;18(4):657-86. doi: 10.1128/CMR.18.4.657-686.2005. PMID 16223952
- [Background] Tamma PD, Rodriguez-Bano J. The Use of Noncarbapenem beta-Lactams for the Treatment of Extended-Spectrum beta-Lactamase Infections. Clin Infect Dis. 2017 Apr 1;64(7):972-980. doi: 10.1093/cid/cix034. PMID 28362938
- [Background] Rodriguez-Bano J, Navarro MD, Retamar P, Picon E, Pascual A; Extended-Spectrum Beta-Lactamases-Red Espanola de Investigacion en Patologia Infecciosa/Grupo de Estudio de Infeccion Hospitalaria Group. beta-Lactam/beta-lactam inhibitor combinations for the treatment of bacteremia due to extended-spectrum beta-lactamase-producing Escherichia coli: a post hoc analysis of prospective cohorts. Clin Infect Dis. 2012 Jan 15;54(2):167-74. doi: 10.1093/cid/cir790. Epub 2011 Nov 4. PMID 22057701
- [Background] Harris PNA, Tambyah PA, Lye DC, Mo Y, Lee TH, Yilmaz M, Alenazi TH, Arabi Y, Falcone M, Bassetti M, Righi E, Rogers BA, Kanj S, Bhally H, Iredell J, Mendelson M, Boyles TH, Looke D, Miyakis S, Walls G, Al Khamis M, Zikri A, Crowe A, Ingram P, Daneman N, Griffin P, Athan E, Lorenc P, Baker P, Roberts L, Beatson SA, Peleg AY, Harris-Brown T, Paterson DL; MERINO Trial Investigators and the Australasian Society for Infectious Disease Clinical Research Network (ASID-CRN). Effect of Piperacillin-Tazobactam vs Meropenem on 30-Day Mortality for Patients With E coli or Klebsiella pneumoniae Bloodstream Infection and Ceftriaxone Resistance: A Randomized Clinical Trial. JAMA. 2018 Sep 11;320(10):984-994. doi: 10.1001/jama.2018.12163. PMID 30208454